CLINICAL TRIAL: NCT01248065
Title: Vitamin D Add-on Therapy Enhances Corticosteroid Responsiveness in Asthma
Brief Title: Study of the Effect of Vitamin D as an Add-on Therapy to Corticosteroids in Asthma
Acronym: VIDA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, dave mauger, Principal Investigator, AsthmaNet Data Coordinating Center, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AsthmaNet 001; 1U10HL098115 (NIH)
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Results first posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-07

CONDITIONS: Asthma
Keywords: Asthma; Vitamin D; Corticosteroids; Treatment failure
MeSH Terms: conditions — Asthma | interventions — Cholecalciferol; ciclesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ciclesonide + placebo (Placebo Comparator)
  Interventions: Drug: Ciclesonide
- Ciclesonide + Vitamin D (Experimental)
  Interventions: Drug: Vitamin D3; Drug: Ciclesonide

INTERVENTIONS:
Drug: Vitamin D3 — vitamin D (100,000 IU loading dose followed by 4,000 IU/day)
  Arms: Ciclesonide + Vitamin D
Drug: Ciclesonide — Low dose inhaled corticosteroid (80 mcg/puff two puffs twice daily)
  Other Names: Alvesco®

SUMMARY:
The purpose of the study is to find out if taking vitamin D in addition to an asthma controller medication helps to prevent worsening of asthma symptoms and asthma attacks.

DETAILED DESCRIPTION:
This is a randomized, double-blind parallel group trial that will enroll individuals who have vitamin D insufficiency and asthma with persistent symptoms despite low-dose inhaled corticosteroid. Participants on low-dose inhaled corticosteroid will be randomized to add-on therapy with either placebo or high-dose vitamin D for a 28-week period. During the inhaled corticosteroid-stable phase, participants will remain on low-dose inhaled corticosteroid. During the inhaled corticosteroid-taper phase, participants will taper their inhaled corticosteroid by 50% at two time-points post-randomization. The investigators will determine if the addition of vitamin D reduces the likelihood of treatment failure when compared to placebo during both the inhaled corticosteroid-stable and inhaled corticosteroid-taper phases of the study. Given the high prevalence of both vitamin D insufficiency and asthma, this trial has high potential to impact daily asthma management.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age and older
* Physician-diagnosed asthma for at least previous 12 months
* Asthma confirmed by: (a) β-agonist reversibility of forced expiratory volume in 1 second (FEV1) ≥12 % following 180 mcg (4 puffs) levalbuterol at visit 1 OR (b) methacholine provocative concentration causing a 20% fall in FEV1 (PC20) ≤ 8 mg/ml if not receiving an inhaled corticosteroid or ≤ 16 mg/ml if receiving an inhaled corticosteroid at visit 2. Source documentation for PC20 from an AsthmaNet methacholine challenge completed within 6 months of visit 2 will be accepted.
* Stable asthma controller therapy (inhaled corticosteroid or leukotriene modifier only) dose for past 2 weeks
* FEV1 ≥ 50% of predicted at visit 1
* Vitamin D level of less than 30 ng/ml at visit 0
* Experienced no more than one treatment failure in the VIDA run-in or oral corticosteroid (OCS) response periods on previous enrollments
* For women of childbearing potential: not pregnant, non-lactating, and agree to practice an adequate birth control method for the duration of the study

Exclusion Criteria:

* Taking vitamin D supplements containing > 1000 IU/day of vitamin D
* Taking >2500 mg/day calcium supplements
* Chronic oral corticosteroid therapy
* Chronic inhaled corticosteroid therapy > 1,000 mcg of fluticasone daily or the equivalent
* History of physician-diagnosed nephrolithiasis
* Use of concomitant medications that alter vitamin D metabolism - phenytoin, phenobarbital, cardiac glycosides; or absorption - orlistat, cholestyramine, colestipol; or those that interfere with study endpoints
* Impaired renal function (GFR < 30 ml/min)
* Asthma exacerbation within past 4 weeks requiring systemic corticosteroids
* Respiratory tract infection within past 4 weeks
* Chronic diseases (other than asthma)
* History of cigarette smoking within the past 1 year or > 10 pack years total
* Serum calcium greater than 10.2 mg/dl on entry
* Urine calcium/creatinine ratio greater than 0.37 (urinary Ca and Creat in mg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2011-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David T. Mauger, PhD, Principal Investigator — Pennsylvania State University College of Medicine; Elliot Israel, MD, Principal Investigator — Brigham and Women's Hospital; Lewis Smith, MD, Principal Investigator — Northwestern Memorial Hospital; Julian Solway, MD, Principal Investigator — University of Chicago; James Moy, MD, Principal Investigator — Rush University Medical Center; Richard Martin, MD, Principal Investigator — National Jewish Health; Christine Sorkness, MD, Principal Investigator — University of Wisconsin, Madison; Elizabeth Bade, MD, Principal Investigator — Aurora Sinai Medical Center; Sally Wenzel, MD, Principal Investigator — University of Pittsburgh Medical Center; James Chmiel, MD, Principal Investigator — Case Western Reserve University School of Medicine; Mario Castro, MD, Principal Investigator — Washington University School of Medicine; Homer Boushey, MD, Principal Investigator — University of California, San Francisco; Monica Kraft, MD, Principal Investigator — Duke University; Stephen Peters, MD, Principal Investigator — Wake Forest University Health Sciences; W. Gerald Teague, MD, Principal Investigator — University of Virginia Health System; Craig LaForce, MD, Principal Investigator — North Carolina Clinical Research; Anne Fitzpatrick, MD, Principal Investigator — Emory University; Jerry Krishnan, MD, Principal Investigator — University of Illinois at Chicago
Locations (16):
- United States (16):
  - University of California - San Francisco, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center/Stroger Hospital, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Duke University School of Medicine, Durham, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Wisconsin-Madison, Madison, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Jiao J, King TS, McKenzie M, Bacharier LB, Dixon AE, Codispoti CD, Dunn RM, Grossman NL, Lugogo NL, Ramratnam SK, Traister RS, Wechsler ME, Castro M; National Heart, Lung, and Blood Institute's AsthmaNet. Vitamin D3 therapy in patients with asthma complicated by sinonasal disease: Secondary analysis of the Vitamin D Add-on Therapy Enhances Corticosteroid Responsiveness in Asthma trial. J Allergy Clin Immunol. 2016 Aug;138(2):589-592.e2. doi: 10.1016/j.jaci.2015.12.1329. Epub 2016 Mar 11. No abstract available. PMID 26971692
- [Derived] Castro M, King TS, Kunselman SJ, Cabana MD, Denlinger L, Holguin F, Kazani SD, Moore WC, Moy J, Sorkness CA, Avila P, Bacharier LB, Bleecker E, Boushey HA, Chmiel J, Fitzpatrick AM, Gentile D, Hundal M, Israel E, Kraft M, Krishnan JA, LaForce C, Lazarus SC, Lemanske R, Lugogo N, Martin RJ, Mauger DT, Naureckas E, Peters SP, Phipatanakul W, Que LG, Sheshadri A, Smith L, Solway J, Sullivan-Vedder L, Sumino K, Wechsler ME, Wenzel S, White SR, Sutherland ER; National Heart, Lung, and Blood Institute's AsthmaNet. Effect of vitamin D3 on asthma treatment failures in adults with symptomatic asthma and lower vitamin D levels: the VIDA randomized clinical trial. JAMA. 2014 May;311(20):2083-91. doi: 10.1001/jama.2014.5052. PMID 24838406

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ciclesonide + Placebo | Ciclesonide + Vitamin D
Started | 207 | 201
Completed | 181 (All 207 participants were included in the primary time-to-event analysis.) | 179 (All 201 participants were included in the primary time-to-event analysis.)
Not Completed | 26 | 22
Not completed — Lost to Follow-up | 3 | 5
Not completed — Withdrawal by Subject | 14 | 11
Not completed — Adverse Event | 3 | 0
Not completed — Third treatment failure event | 3 | 1
Not completed — Other | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciclesonide + Placebo | Ciclesonide + Vitamin D | Total
Number analyzed (Participants) | 207 | 201 | 408
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (12.7) | 39.9 (13.1) | 39.7 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 137 | 278
  Male | 66 | 64 | 130
Race/Ethnicity, Customized [Number; unit: participants]
  Asian/Pacific Islander | 7 | 7 | 14
  Black | 68 | 63 | 131
  White | 111 | 105 | 216
  Hispanic | 19 | 20 | 39
  Other | 2 | 6 | 8
Duration of asthma [Mean (Standard Deviation); unit: years] | 25.0 (12.8) | 24.9 (13.5) | 25.0 (13.2)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 31.5 (9.5) | 32.0 (8.2) | 31.8 (8.9)
Symptom score (morning) [Mean (Standard Deviation); unit: Avg score of 5 sx: 0=absent to 3=severe] | 0.41 (0.36) | 0.41 (0.34) | 0.41 (0.35)
Symptom score (afternoon and evening) [Mean (Standard Deviation); unit: Avg score of 5 sx: 0=absent to 3=severe] | 0.43 (0.40) | 0.44 (0.35) | 0.43 (0.37)
Level of 25-hydroxyvitamin D [Median (Inter-Quartile Range); unit: ng/mL] | 18.8 [13.4 to 23.7] | 19.9 [14.5 to 25.0] | 19.2 [13.9 to 24.3]
FEV1 before albuterol use (L) [Mean (Standard Deviation); unit: liters] | 2.62 (0.83) | 2.63 (0.78) | 2.63 (0.80)
FEV1 before albuterol use (% predicted) [Mean (Standard Deviation); unit: % predicted] | 80.5 (14.2) | 80.7 (13.8) | 80.6 (14.0)
Methacholine PC20 (mg/mL) [Geometric Mean (Standard Deviation); unit: mg/mL] | 1.85 (1.67) | 2.05 (1.61) | 1.95 (1.65)
Sputum eosinophils (%) [Median (Inter-Quartile Range); unit: % of eosinophils] | 0.40 [0 to 1.30] | 0.30 [0 to 1.30] | 0.40 [0 to 1.30]

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure
Description: Treatment failure is a well-defined asthma outcome reflecting overall asthma control that has been used previously in multiple clinical trials. Treatment failure as defined in the current proposal and prior trials is consistent with the American Thoracic Society (ATS)/European Respiratory Society(ERS) definition of a moderate exacerbation - a deterioration in symptoms and/or lung function with increased rescue bronchodilator use that lasts 2 days or more. The percentages of participants experiencing a treatment failure are Kaplan-Meier estimates of failure rate.
Time Frame: Twenty-eight week intervention period from randomization until end of trial.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ciclesonide + Placebo | Ciclesonide + Vitamin D
Number analyzed (Participants) | 207 | 201
Percentage of participants | 29 [23 to 35] | 28 [21 to 34]

2. Secondary Outcome: Lung Function Change From Baseline
Description: FEV1 (liters) and methacholine PC20 will be evaluated. Changes are measured as 28 weeks minus baseline.
Time Frame: Change is measured as value at 28 weeks minus baseline value.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Ciclesonide + Placebo | Ciclesonide + Vitamin D
Number analyzed (Participants) | 207 | 201
Liters | -0.04 [-0.11 to 0.03] | -0.07 [-0.14 to 0.01]

3. Secondary Outcome: Exacerbations
Description: Outcome defined as number of exacerbations per person-year.
Time Frame: Overall exacerbation rate during 28-week trial
Measure: Number (95% Confidence Interval); unit: Exacerbations/person-year
Arm/Group | Ciclesonide + Placebo | Ciclesonide + Vitamin D
Number analyzed (Participants) | 207 | 201
Exacerbations/person-year | 0.40 [0.30 to 0.50] | 0.26 [0.18 to 0.33]

ADVERSE EVENTS:
Arm/Group | Ciclesonide + Placebo | Ciclesonide + Vitamin D
Serious Adverse Events (participants affected / at risk) | 9/207 | 6/201
Other Adverse Events (participants affected / at risk) | 157/207 | 168/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciclesonide + Placebo (N=207) | Ciclesonide + Vitamin D (N=201)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 1 (1)
Initial diagnosis of breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Severe leg pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sigmoid diverticulitis with abscess (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastric volvulus causing gastric outlet obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Major depression disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Allergic reaction/rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Benign fibroid tumor surgery (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Inguinal hernia (Surgical and medical procedures) | 0 (0) | 1 (1)
Transient ischemic attack (General disorders) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Limb edema (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ciclesonide + Placebo (N=207) | Ciclesonide + Vitamin D (N=201)
Diseases of the digestive system (Gastrointestinal disorders) | 23 (28) | 13 (20)
Diseases of the genitourinary system (Renal and urinary disorders) | 18 (31) | 12 (12)
Diseases of the musculoskeletal system and connective tissue (Musculoskeletal and connective tissue disorders) | 31 (46) | 29 (33)
Diseases of the nervous system and sense organs (Nervous system disorders) | 25 (27) | 23 (30)
Diseases of the respiratory system (Respiratory, thoracic and mediastinal disorders) | 122 (231) | 137 (253)
Infectious and parasitic diseases (Infections and infestations) | 22 (23) | 12 (13)
Injury and poisoning (Injury, poisoning and procedural complications) | 23 (31) | 28 (40)
Symptoms, signs, and ill-defined conditions (General disorders) | 60 (114) | 59 (141)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No